CLINICAL TRIAL: NCT00841750
Title: The NoTube Study: Evaluation of the Necessity of a Chest Tube After a Video-assisted Thoracoscopic Surgery Pulmonary Wedge Resection.
Brief Title: Chest Tube After a Video-assisted Thoracoscopic Surgery Pulmonary Wedge Resection
Acronym: NOTUBE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle (Other)
Collaborators: Universidad Industrial de Santander (Other); Clinica Chicamocha (Unknown)
Responsible Party: Leonidas Tapias Diaz, Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9009001
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Lung Diseases, Interstitial; Pulmonary Nodule, Solitary
Keywords: Chest Tubes; Thoracic Surgery, Video-Assisted; Lung Diseases, Interstitial; Pulmonary Nodule, Solitary
MeSH Terms: conditions — Lung Diseases, Interstitial; Solitary Pulmonary Nodule

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No chest tube (Experimental): No chest tube left in the pleural cavity at the end of a VATS pulmonary wedge resection.
  Interventions: Procedure: Do not leave a chest tube in the pleural cavity.
- Chest tube (Active Comparator): Chest tube left in the pleural cavity at the end of a VATS pulmonary wedge resection.
  Interventions: Procedure: Do leave a chest tube in the pleural cavity.

INTERVENTIONS:
Procedure: Do not leave a chest tube in the pleural cavity. — At the end of a VATS wedge resection, an air leak proof will take place and if no air leak is noted, the surgical incisions for thoracoscopy ports will be closed without leaving a chest tube inserted in the pleural cavity of the patient.
  Arms: No chest tube
Procedure: Do leave a chest tube in the pleural cavity. — At the end of a VATS wedge resection, a chest tube will be inserted in the pleural cavity of the patient through the inferior surgical incision for thoracoscopy port; the rest of the incisions will be closed.
  Arms: Chest tube

SUMMARY:
After performing VATS pulmonary wedge resections, a chest tube is routinely left in the pleural cavity to drain possible air leaks and fluid accumulations. Chest tubes after VATS pulmonary wedge resections are left in place a minimum of 1 day. However, this practice has no scientific foundations. The investigators believe it is possible to avoid the placement of a chest tube after this procedure in a great amount of patients. This is a randomized controlled clinical trial with analysis blinding in which the investigators want to compare the outcomes between installing a chest tube or not after VATS pulmonary wedge resections. The investigators will include consecutively patients with interstitial lung disease or indeterminate pulmonary nodules undergoing this procedure, at the participating institutions. The investigators calculated a sample size of 50 subjects in each group using pneumothorax < 10% data from Luckraz et al and to determine a difference of hospital stay of 2 versus 1 day; DS(1.5), power = 0.9 and alpha = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing video-assisted thoracoscopic surgery pulmonary wedge resections at the participating institutions.
* No evidence of air leak at the end of the surgical procedure.
* No active bleeding at the end of the surgical procedure.

Exclusion Criteria:

* Pleural effusion previous to the procedure requiring drainage after it.
* Bullous or emphysematous changes in lung parenchyma.
* Patients going to positive pressure in the airways after the procedure.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Pneumothorax >10% / Hemothorax | 1 hour and 1-5 days postoperatively

SECONDARY OUTCOMES:
Pain (Visual analogue scale) | At days 1-5 of hospitalization and at 1 month
Surgical procedure duration | At the end of surgery
Hospital stay | At patient discharge

CONTACTS AND LOCATIONS:
Overall Officials: Leonidas Tapias, MD, Principal Investigator — Fundacion Oftalmológica de Santander Clinica Carlos Ardila Lulle; Luis C Orozco-Vargas, MD, Principal Investigator — Universidad Industrial de Santander; Luis F Tapias-Vargas, Study Chair — Universidad Industrial de Santander
Locations (3):
- Colombia (3):
  - Fundacion Santa Fe de Bogota, Bogotá, Bogota D.C.
  - Clinica Chicamocha, Bucaramanga, Santander Department
  - Fundacion Oftalmológica de Santander Clinica Carlos Ardila Lulle, Floridablanca, Santander Department